CLINICAL TRIAL: NCT03961217
Title: Return to Work Among Cancer Survivors With Treatment-induced Survivorship Syndromes
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Gunnar Steineck, Professor / Senior consultant, Sahlgrenska University Hospital
Other Study IDs: ANB_691-17
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Gynecologic Cancer; Prostate Cancer; Radiation Toxicity; Malignancy; Radiotherapy Side Effect; Radiation Injuries; Cancer Survivors; Radiation Syndrome
Keywords: Return to work; Disability pension; Sickness Absence; Employability; Fitness to work; Wellbeing; Radiotherapy Side Effect; Cancer Survivors
MeSH Terms: conditions — Prostatic Neoplasms; Radiation Injuries; Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Gynecological Cases: Gynecological Cancer survivors with treatment induced survivorship syndroms treated pelvic radiotherapy at
  1. Radiumhemmat, Karolinska University Hospital and
  2. Jubileumskliniken at Sahlgrenska University Hospital in Sweden.
  Interventions: Radiation: Radiotherapy
- Prostate Cases: Prostate Cancer survivors treated with radiotherapy for localized prostate cancer at Sahlgrenska University Hospital, Gothenburg, Sweden
  Interventions: Radiation: Radiotherapy
- Gynecological Rehab Cases: Gynecological Cancer survivors with treatment induced survivorship syndroms treated pelvic radiotherapy
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy as part of cancer treatment

SUMMARY:
The investigators plan to investigate the consequences of late effects (radiation-induced survivorship syndromes) after radiotherapy in Gynecological and Prostate cancer survivors on return to work (Yes/No) and if RTW happened then time to RTW.

In addition, whether general health, type of work (occupation), work environment factors, individual factors (lifestyle, socioeconomic status etc.), contribute to the adverse late effects of radiotherapy and these Gynecological cancer survivors have a higher risk for disability pension/long term sickness absence (NOT Return to work).

DETAILED DESCRIPTION:
Occurrence of cancer diagnoses are rising, and both disease and treatments are aggressive. Due to advancement in medical technology, improved therapy and/or early detection the overall survival rates are also improving.

Some of the most common cancer types, such as breast cancer, prostate cancer, cervical cancer, and colorectal cancer have high cure rates when detected early and treated according to best practices. Many of these cancer survivors are of working age and are likely to return to work. Women who survive cervical cancer and men who survive testicular cancer typically have three to four decades left in working life.

However, return to work (RTW) among cancer survivors may not be similar to RTW among long-term sickness absentees due to other diagnoses. Cancer is a life threatening disease and cancer diagnose is a life changing event. The emotional shock after the cancer diagnosis may be associated with low psychological well-being even two years after prostate cancer surgery.

The successful cancer treatment concludes with the lifelong consequences of surgery, irradiation, cytotoxic chemotherapy, biological anticancer substances or other drugs in the treatment. The ionizing radiation that eliminates malignant cells may trigger long-lasting pathophysiological processes in the normal tissue and affect the health of the survivors with lifelong treatment-induced survivorship diseases. In a recent study, Steineck et al, identified five radiation-induced survivorship syndromes affecting bowel health in a cohort of gynecological cancer; urgency syndrome (30%), leakage syndrome (26%), excessive gas discharge(15%), excessive mucus discharge (16%) and blood discharge (10%).

There is a lack of knowledge about how these side effects of cancer treatment affect the degree of work ability and return to work. Clinical experience suggests that many cancer survivors have reduced work ability. There is a need for scientific studies that shed light on the side effects of cancer treatment and their relation to work ability.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25 to 60 years (working age)
2. Employed at time of diagnosis
3. Treated for cancer
4. Suffering from at least one of Radiation-induced survivorship syndromes
5. First cancer & first time treatment for cancer,

Exclusion Criteria:

1. No other chronic disease
2. Chronic intestinal illness/surgery
3. Stage IV cancer
4. Recurrent cancer/Relapse

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Gyaecological cancer survivors Prostate cancer survivors
Study Population: Cohort of women treated with external pelvic radiotherapy for a gynaecological malignancy and men treated with radiotherapy for prostate cancer at two large oncology clinics in Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 2135 (Actual)
Dates: Start 1991-01 (Actual); Primary Completion 2006-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Return to work (RTW) | Five - Ten years after mapping Radiation-induced survivorship syndromes
  Information on Sickness absence for more than 14 days was obtained from the official registries in Sweden.

SECONDARY OUTCOMES:
Time to Return to work | Five - Ten years after mapping Radiation-induced survivorship syndromes
  Sickness absence (more than 14 days) until the survivor returned to work. Also obtained from the official registries in Sweden.

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Steineck, Principal Investigator — Clinical Cancer Epidemiology, Sahlgrenska Academy, Gothenburg, Sweden
Locations (1):
- Jubileumskliniken, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steineck G, Skokic V, Sjoberg F, Bull C, Alevronta E, Dunberger G, Bergmark K, Wilderang U, Oh JH, Deasy JO, Jornsten R. Identifying radiation-induced survivorship syndromes affecting bowel health in a cohort of gynecological cancer survivors. PLoS One. 2017 Feb 3;12(2):e0171461. doi: 10.1371/journal.pone.0171461. eCollection 2017. PMID 28158314
- [Background] Dunberger G, Lind H, Steineck G, Waldenstrom AC, Nyberg T, Al-Abany M, Nyberg U, Vall-Lundqvist E. Self-reported symptoms of faecal incontinence among long-term gynaecological cancer survivors and population-based controls. Eur J Cancer. 2010 Feb;46(3):606-15. doi: 10.1016/j.ejca.2009.10.023. Epub 2009 Nov 18. PMID 19926277
- [Background] Alsadius D, Hedelin M, Johansson KA, Pettersson N, Wilderang U, Lundstedt D, Steineck G. Tobacco smoking and long-lasting symptoms from the bowel and the anal-sphincter region after radiotherapy for prostate cancer. Radiother Oncol. 2011 Dec;101(3):495-501. doi: 10.1016/j.radonc.2011.06.010. Epub 2011 Jul 5. PMID 21737169
- [Background] Lind H, Waldenstrom AC, Dunberger G, al-Abany M, Alevronta E, Johansson KA, Olsson C, Nyberg T, Wilderang U, Steineck G, Avall-Lundqvist E. Late symptoms in long-term gynaecological cancer survivors after radiation therapy: a population-based cohort study. Br J Cancer. 2011 Sep 6;105(6):737-45. doi: 10.1038/bjc.2011.315. Epub 2011 Aug 16. PMID 21847122
- [Derived] Noor Baloch A, Hagberg M, Thomee S, Steineck G, Sanden H. The physical and psychological aspects of quality of life mediates the effect of radiation-induced urgency syndrome on disability pension in gynecological cancer survivors. Cancer Med. 2023 Aug;12(16):17377-17388. doi: 10.1002/cam4.6356. Epub 2023 Jul 24. PMID 37489096
- [Derived] Baloch AN, Hagberg M, Thomee S, Steineck G, Sanden H. Disability pension among gynaecological cancer survivors with or without radiation-induced survivorship syndromes. J Cancer Surviv. 2022 Aug;16(4):834-843. doi: 10.1007/s11764-021-01077-9. Epub 2021 Aug 19. PMID 34414517
- See also: Self-reported symptoms of faecal incontinence among long-term gynaecological cancer survivors and population-based controls — https://doi.org/10.1016/j.ejca.2009.10.023
- See also: Identifying radiation-induced survivorship syndromes affecting bowel health in a cohort of gynecological cancer survivors — https://dx.doi.org/10.1371%2Fjournal.pone.0171461
- See also: Tobacco smoking and long-lasting symptoms from the bowel and the anal-sphincter region after radiotherapy for prostate cancer — https://doi.org/10.1016/j.radonc.2011.06.010
- See also: Late symptoms in long-term gynaecological cancer survivors after radiation therapy: a population-based cohort study — https://www.nature.com/articles/bjc2011315